CLINICAL TRIAL: NCT03212040
Title: Comparison of Needle Gauge 14 vs. Gauge 16 in Breast Biopsy
Brief Title: 14 g vs. 16 g in Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Gauge 14/16
Record Dates: First submitted 2017-06-27; First posted 2017-07-11 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2019-02

CONDITIONS: Breast Biopsy
MeSH Terms: interventions — Biopsy, Needle

STUDY DESIGN:
Intervention Model Description: Comparison of 14 vs 16 gauge needles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14 gauge needle biopsy (Active Comparator): breast biopsy will be performed with 14 gauge needle
  Interventions: Diagnostic Test: needle biopsy
- 16 gauge needle biopsy (Active Comparator): breast biopsy will be performed with 16 gauge needle
  Interventions: Diagnostic Test: needle biopsy

INTERVENTIONS:
Diagnostic Test: needle biopsy — breast biopsy using different needle gauges

SUMMARY:
Comparison of biopsy needles with a different diameter, i.e. 14 vs 16 gauge, used for breast biopsies

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Informed consent available
* Palpable and non-palpable breast findings
* Tumor size 5-20 mm
* Findings of sonographic BI-RADS® classification 2-5.
* Guideline-oriented indication for bioptic clarification

Exclusion Criteria:

* No reliable sonographic demarcation of the finding
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2013-02-18 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  * Diagnostic aggreement (representativity) with definitive histology of core needle specimen and of surgical specimen
  * Additive diagnostic aggreement (representativity) with definitive histology of core needle specimen and with histology of surgical specimen, with 1 to 5 passes of core needle biopsy
  * Additive diagnostic accuracy to achieve a high (>=99%) diagnostic yield, with 1-5 passes of core needle biopsy
Diagnostic quality | 1 year
  * Diagnostic quality of specimen to achieve an accurate histological diagnosis
  * Diagnostic quality of specimen to achieve an accurate histological diagnosis, with 1 to 5 passes of core needle biopsy
  * Additive diagnostic quality to achieve a high (>=99%) diagnostic yield, with 1-5 passes of core needle biopsy

SECONDARY OUTCOMES:
Pain related to the biopsy procedure | 1 year
  Subjective pain perception measured visual analog scale
Duration time of the biopsy procedure | 1 year
  Duration time of the biopsy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No